CLINICAL TRIAL: NCT06149481
Title: Phase I/II Study of the Combination Immunotherapy Regimen: SX-682, TriAdeno Vaccine, Retifanlimab and IL-15 Agonist N-803 (STAR15) for Metastatic Colorectal Cancer (mCRC)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 10001563; 001563-C
Record Dates: First submitted 2023-11-28; First posted 2023-11-29 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-11-18

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Monoclonal Antibody; Brachyury; MUC-1; Immunoglobulin G cytokine fusion protein; chemokine antagonist; Small Molecule
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Brachyury Protein; ALT-803

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Retifanlimab + TriAdeno Vaccine + N-803
  Interventions: Drug: Retifanlimab; Biological: Therapeutic CEA, Brachyury and MUC1 TriAdeno Vaccine Platform; Drug: N-803
- Arm 2 (Experimental): Retifanlimab + TriAdeno Vaccine + N-803 + SX-682
  Interventions: Drug: Retifanlimab; Biological: Therapeutic CEA, Brachyury and MUC1 TriAdeno Vaccine Platform; Drug: N-803; Drug: SX-682

INTERVENTIONS:
Drug: Retifanlimab — 500 mg infused via IV over 30 minutes every 28 days
Biological: Therapeutic CEA, Brachyury and MUC1 TriAdeno Vaccine Platform — 5x10^11 virus particles per 1 mL administered via subcutaneous injection in the upper arm and anterolateral upper thigh on Day 1 of Cycles 1, 2, 3 and every 3 cycles after that
Drug: N-803 — 15 ug/kg administered via subcutaneous injection to the abdomen every 28 days
Drug: SX-682 — 100 mg administered orally twice per day on days 6-26 of every cycle
  Arms: Arm 2

SUMMARY:
Background:

Each year, more than 32,000 people in the United States are diagnosed with colorectal cancer that has returned or progressed after treatment and spread to other organs. This is called metastatic colorectal cancer (mCRC). Most people with mCRC survive only about 2 years.

Objective:

To test the ability of a combination of up to 4 experimental anti-cancer drugs treat mCRC. The names of these drugs are retifanlimab, TriAdeno vaccine, N-803, and SX-682. They are described below.

Eligibility:

Adults aged 18 years or older with mCRC. Participants must have

Design:

Participants will be screened. This includes having a physical exam, blood tests, urine tests, and imaging tests. If signed on to the study, participants will have 2 tumor biopsies. One when starting the study and once about 8 weeks after bring on the study. Participants will receive $500 for each biopsy.

Participants will be treated with either 3 or 4 drugs and will receive a detailed calendar explaining when each drug is given.

Retifanlimab is given every 4 weeks through an IV (an IV is tube attached to a needle inserted into a vein in the arm). N-803 is injected under the skin on the abdomen every 4 weeks.

TriAdeno vaccine is injected under the skin of the upper arm or thigh once a month for 3 doses and then once every 3 months.

Some participants will also receive a 4th drug. SX-682 is a pill taken by mouth. Participants will take this drug 2 times a day at home for about 3 weeks of each month.

Study treatment will continue up to 2 years. Follow-up phone calls/emails may continue for 3 more years.

DETAILED DESCRIPTION:
Background:

* mCRC is incurable and available standard therapies offer a median overall survival of approximately 2 years.
* Most cases (approximately 95%) of mCRC have an intact expression of DNA mismatch repair enzymes (MLH1, MSH2, MSH6, and PMS2), and are commonly classified as having mismatch repair proficient (pMMR) or microsatellite stable (MSS) mCRC.
* MSS mCRC does not respond to immune checkpoint inhibitor (ICI) therapy whereas mismatch repair deficient (or microsatellite instability-high) mCRC is responsive to ICI therapy.
* Preclinical and clinical studies conducted at the NCI in the Laboratory of Tumor Immunology Biology (LTIB) indicate that the combination of programmed cell death protein 1 (PD-1) / Programmed death-ligand 1 (PD-L1) blockade, tumor-associated antigens (TAA) targeted vaccine, IL15 agonist, and CXCR1/2 inhibition may include sufficient immune enhancements to produce anti-tumor activity in MSS mCRC.
* Retifanlimab is a humanized IgG4 monoclonal antibody that targets PD-1. Retifanlimab has been studied in several clinical trials, and several malignancies, and has a safety and clinical activity profile similar to approved anti-PD-1 therapies (e.g., pembrolizumab).
* The TriAdeno Vaccine employs 3 adenovirus serotype 5 vectors, encoding three TAAs (CEA, MUC1, and brachyury). These vaccines have completed the phase 1 study and are safe and well tolerated. Vaccination generates antigen-specific T cell responses to CEA, MUC1, and brachyury.
* N-803 is an IL-15 agonist that activates and expands T cells and NK cells. N-803 enhances anti-tumor activity in combination with tumor-targeted vaccines. Clinically, multiple studies have demonstrated the safety of tumor-targeted vaccine in combination with PD- 1/PD-L1 blockade. Adding N-803 to PD-1/PD-L1 blockade can produce antitumor responses in disease states where responses to PD-1/PD-L1 alone would not be expected.
* SX-682 is a small molecule, orally bioavailable, allosteric antagonist of the chemokine receptors CXCR1 and CXCR2. Inhibition of CXCR1 and CXCR2 addresses a major component of intratumoral T cell suppression by myeloid-derived suppressor cells and tumor-associate macrophages. SX-682 has shown to be tolerable in combination with PD- 1/PD-L1 blockade.

Objectives:

* Phase I: to describe the safety profile of the Immuno-Oncology (IO) regimens consisting of retifanlimab, TriAdeno vaccine, N-803 (A1), and retifanlimab, TriAdeno vaccine, N- 803, SX 682 (A2) in participants with metastatic colorectal cancer (mCRC).
* Phase II: to determine the objective response rate (ORR) (complete response (CR) + partial response (PR)) of the IO regimen in mCRC.

Eligibility:

* Age >=18 years.
* Previously treated metastatic colorectal cancer with measurable disease.
* Eastern Cooperative Oncology Group (ECOG) performance status <= 2.
* Adequate organ function.

Design:

* This is an open-label Phase I/II trial to evaluate the safety and efficacy of the Immuno- Oncology regimen, consisting of retifanlimab, TriAdeno vaccine, N-803, and SX-682 in participants with mCRC.
* During Phase I, we will assess the safety of the three- and the four-drug IO regimens.
* During Phase II we will continue to evaluate the safety and examine the efficacy of the four drug IO regimen. If 0 to 1 of the first 9 participants treated with the 4-drug IO regimen have a clinical response, defined as complete response (CR) + partial response (PR) within the first 24 weeks after treatment initiation, then no further participants will be accrued using the quadruple combination. If 2 or more of the first 9 participants have a response, then accrual will continue until a total of 23 evaluable participants have been treated with a four-drug IO regimen.
* Participants will receive treatment in cycles consisting of 28 (+7) days for 2 years.
* To allow for a small number of inevaluable participants, and screen failures the accrual ceiling will be set at 60.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Participants with histologically confirmed colorectal cancer and evidence of metastatic disease.
* Participants must have received, been ineligible to receive, or refused to receive two lines of standard systemic therapy i.e., a fluoropyrimidine with oxaliplatin or irinotecan with bevacizumab, regorafenib, trifluridine, and (if history of RAS wild-type) EGFR-targeted therapy. Participants must have received one line of systemic checkpoint inhibitor if history of advanced microsatellite instability-high [MSI-H/dMMR]) metastatic colon cancer.
* Participants who had progressive disease within 6 months before study treatment following standard adjuvant therapy are eligible if they have not received systemic therapy for metastatic disease. Participants with a history of MSI-H/dMMR must have also received one line of checkpoint inhibitor therapy.
* Age >= 18 years.
* Measurable disease per RECIST 1.1.
* ECOG performance status <= 2.
* Adequate organ and marrow as a function defined below:

  * absolute neutrophil count (ANC) >= 1,500 cells/mm^3
  * platelet count >= 100,000 cells/mm^3
  * hemoglobin (Hgb) >= 9 g/dL
  * total bilirubin level < 1.5 x upper limit of normal (ULN)
  * alanine aminotransferase (ALT) <= 2.5 x ULN OR <= 5 x ULN for participants with liver metastases
  * aspartate aminotransferase (AST) level <= 2.5 x ULN OR <= 5 x ULN for participants with liver metastases
  * creatinine clearance (CrCl) calculated by Cockroft-Gault formula >= 50 mL/min
* Resolution of toxic effect(s) of prior anti-cancer therapy (except alopecia and neuropathy) to Grade <=1 or to <=2 if effective medical management of those toxicities is in place such that they are controlled per standard of care (e.g., grade 2 hypothyroidism requiring oral thyroid replacement).
* Participants with treated brain metastases are eligible if clinically appropriate follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression.
* Participants positive for human immunodeficiency virus (HIV) are eligible if they are compliant with appropriate anti-retroviral therapy for at least 6 months, have HIV viral load <400 copies/mL, and a CD4 count > 350 cells/microliter at screening.
* Participants positive for Hepatitis C virus (HCV) are eligible if they have completed definitive anti-viral therapy and have an undetectable viral load.
* Individuals of child-bearing potential (IOCBP) and individuals who can father children must agree to use an effective method of contraception (barrier, hormonal, intrauterine device [IUD], surgical sterilization) at study entry and up to 6 months after the last dose of the study drug(s).
* Breastfeeding participants must be willing to discontinue breastfeeding from study treatment initiation through 6 months after study treatment discontinuation.
* Participants must have lesion(s) accessible for biopsy (other than used for measurement of disease) and be willing to undergo mandatory study biopsies. Lesions to be biopsied will be determined safely accessible by the provider performing the biopsy (e.g. interventional radiology if a liver or lung biopsy) prior to performing the biopsy.
* Participants must be able to understand and willing to sign a written informed consent document.

EXCLUSION CRITERIA:

* Participants with prior investigational drug, chemotherapy, immunotherapy, or any prior therapeutic radiotherapy within 14 days prior to study treatment initiation.
* Participants with palliative radiotherapy performed within 7 days prior to study treatment initiation.
* Active autoimmune disease requiring systemic immunosuppression in excess of physiologic maintenance doses of corticosteroids (> 10 mg/day of prednisone or equivalent) with the exception of:

  * intermittent use of bronchodilators, inhaled corticosteroids, or local corticosteroid injections in participants with asthma
  * using topical, ocular, intra-articular, or intranasal corticosteroids (with minimal systemic absorption
  * brief courses of corticosteroids for prophylaxis (e.g., contrast dye allergy).
* Evidence of interstitial lung disease, history of interstitial lung disease, or active, noninfectious pneumonitis. Participants with chronic post-radiation pulmonary changes/scarring that is asymptomatic are eligible.
* Active infections requiring systemic antibiotics or antifungal or antiviral treatment within 8 days prior to treatment initiation. Participants who have had appropriate antibiotics initiated but are still completing the treatment course are eligible if clinically improved or had minimal symptoms at presentation (e.g., urinary tract infection or pharyngeal streptococcal infection without evidence of systemic inflammatory response).

  * History of organ transplant, including allogeneic stem cell transplantation.
  * Participants who experienced immune-related toxicity during prior checkpoint inhibitor therapy for which permanent discontinuation of therapy was recommended (per product label or consensus guidelines) or any immune-related toxicity requiring systemic corticosteroids (with the exception of endocrinopathy that is well controlled on replacement hormones).
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to the study drugs.
* Receipt of a live vaccine within 28 days prior to treatment initiation. Note: Examples of live vaccines include but are not limited to measles, mumps, rubella, varicella-zoster (chickenpox), yellow fever, rabies, BCG, and typhoid vaccines. Seasonal influenza vaccines for injection are generally killed-virus vaccines and are allowed; however, intranasal influenza vaccines are live, attenuated vaccines and are not allowed.
* History of infection with Hepatitis B virus (HBV) unless on suppressive therapy. Individuals with serologic evidence of a resolved prior HBV infection (i.e., HBsAgnegative and anti-HBc positive) are eligible.
* Pregnancy confirmed with Beta-human chorionic gonadotropin (Beta-HCG) serum or urine pregnancy test performed in IOCBP at screening.
* Uncontrolled intercurrent illness that would limit compliance with study requirements.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-03-26 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2030-10-31 (Estimated)

PRIMARY OUTCOMES:
Phase I: Safety profiles of the IO regimens consisting of retifanlimab, TriAdeno vaccine, N-803 (A1), and retifanlimab, TriAdeno vaccine, N-803, SX-682 (A2) in participants with metastatic colorectal cancer | Day 1 of Cycle 1 through 30 days after the last study drug administration
  Number of DLTs within DLT period (C1 days 1-28). Any toxicities identified.
Phase II: Overall response rate (ORR) defined as the CR+PR of the IO regimen in mCRC | Every 8 weeks until either disease progression or 2 years after initiation of study therapy.
  The fraction of participants with a CR or PR (per RECIST v1.1) in Phase II will be reported along with a 95% confidence interval.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) at 6, 12, and 24 months | Every 8 weeks until disease progression or for 2 years after initiation of study therapy
  PFS will be determined by the Kaplan-Meier method and reported at 6, 12, and 24 months from the date the participant was enrolled in the trial, along with 95 percent confidence intervals at these times.
Disease control rate (DCR) at 6 and 12 months | Every 8 weeks until disease progression or 1 year after initiation of study therapy
  DCR at 6 and 12 months will be reported as a fraction along with a 95 percent confidence interval for each.
Safety during Phase II | From Day 1 to 30 days of the last study drug administration
  AEs will be reported by type and grade within Phase II.
Overall survival | Up to 2 years after start of study therapy
  Monitoring of participants from Day 1 of each cycle, at follow up visits and until date of death/closure of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas P Tschernia, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD will be shared. All IPD recorded in the medical record will be shared with intramural investigators upon request. In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data from this study may be requested from other researchers within 10 years after the completion of the primary endpoint. Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Data from this study may be requested by contacting the PI. Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001563-C.html